CLINICAL TRIAL: NCT02641821
Title: Effect of Nifedipine GITS in Patients With Mild-to-moderate Primary Hypertension: a Multi-center, Open-label, Observational Study
Brief Title: Effect of Nifedipine GITS in Patients With Mild-to-moderate Primary Hypertension
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking University First Hospital (Other)
Collaborators: Bayer (Industry)
Responsible Party: Principal Investigator, Yong Huo, Director, Department of Cardiology, Peking University First Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Nifedipine-HT-1.0
Record Dates: First submitted 2015-12-18; First posted 2015-12-29 (Estimated); Last update posted 2019-03-22 (Actual); Status verified 2019-03

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Nifedipine GITS (Experimental)
  Interventions: Drug: Nifedipine GITS

INTERVENTIONS:
Drug: Nifedipine GITS

SUMMARY:
This is a multi-center, open-label, observational study. The aim of this study is to evaluate the efficacy of Nifedipine GITS on lowering blood pressure in Chinese adults with mild-to-moderate hypertension.

DETAILED DESCRIPTION:
The primary aim of the study is to evaluate the efficacy of nifedipine gastrointestinal therapeutic system (GITS) on lowering blood pressure in Chinese adults with mild-to-moderate hypertension. The secondary aim of the study is to evaluate the efficacy of Nifedipine GITS on lowering blood pressure in hypertensive patients with different urinary sodium levels. Based on sample size estimation, the plan is to recruit 700 patients from 16 centers. At baseline, patients'demographic characters, disease history and anthropometric indices will be collected, laboratory tests will be performed for blood routine examination, urinalysis, renal function, hepatic function, urinary sodium and 24-hour urinary sodium. All eligible patients will be assigned to a treatment of Nifedipine GITS and followed up for 8 weeks. At 0 day, 2,weeks, 4 weeks and 8 weeks of the study, seated blood pressure, vital signs, medication and adverse events were collected. At the end of the study, 24-hour ambulatory blood pressure monitoring (ABPM) will be performed for all participants.

ELIGIBILITY:
Inclusion Criteria:

* a seated systolic BP (SBP) ≥140 mmHg and <180 mmHg and/or a seated diastolic BP (DBP) ≥90 mmHg and <110 mmHg;
* an age ≥18 and ≤75 years;
* those who had not taken any BP-lowering medications in 1 month before the study.

Exclusion Criteria:

* a seated systolic BP (SBP) ≥180 mmHg and/or a seated diastolic BP ≥110 mmHg;
* secondary hypertension;
* diagnosed heart failure or stroke;
* Any of alanine aminotransferase (ALT) or aspartate aminotransferase (AST) was above 1.5 times of it's normal value upper limit, Serum creatinine >177 µmmol/L (2mg/dL), or liver cirrhosis;
* subjects with carotid stenosis or systolic murmur
* subjects with a history of unstable angina pectoris, acute mycardial infarction, percutaneous transluminal coronary angiography or coronary artery bypass grafting in the past 6 months;
* subjects who were within lactation period, pregnant, or planning to become pregnant during the study;
* hypersensitive to Nifedipine GITS or with SAE;
* subjects who are participating in other clinical trials;
* considered not fit for the study due to other reasons according to the researchers (such as Malignant tumor, psyche or nervous system dysfunction, or special diseases).

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 700 (Estimated)
Dates: Start 2015-10; Primary Completion 2019-12 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Control rate of hypertension evaluated by office blood pressure at 8 weeks | 8 weeks
Control rate of hypertension evaluated by office blood pressure at 4 weeks | 4 weeks
Control rate of hypertension evaluated by office blood pressure at 2 weeks | 2 weeks

SECONDARY OUTCOMES:
Control rate of hypertension evaluated by 24-hour ABPM at 8 weeks | 8 weeks
Change of office blood pressure from baseline to 8 weeks | 8 weeks
Change of 24-hour ABPM from baseline to 8 weeks | 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Yong Huo, MD, Principal Investigator — Peking University First Hospital
Locations (1):
- Division of Cardiology, Peking University First Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: Undecided